CLINICAL TRIAL: NCT00120861
Title: A Randomized, Phase IIb Clinical Trial to Evaluate the Safety and Antiviral Activity of NM283 and the Combination of Pegylated Interferon Plus NM283, in Patients With Chronic Hepatitis C Who Have Previously Failed to Respond to Standard Therapy
Brief Title: Valopicitabine Alone and Together With Pegylated Interferon in Patients With Chronic Hepatitis C Who Have Failed to Respond to Standard Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV-08A-004
Record Dates: First submitted 2005-07-11; First posted 2005-07-19 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis C
Keywords: Genotype-1; Previously failed treatment
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — valopicitabine; Ribavirin

INTERVENTIONS:
Drug: valopicitabine
Drug: pegylated interferon
Drug: ribavirin

SUMMARY:
This study is being conducted to compare the safety, effectiveness and tolerance of valopicitabine (NM283) when used alone and when valopicitabine is used together with pegylated interferon in hepatitis C treatment failure patients. These results will be compared against the results of treatment with pegylated interferon plus ribavirin, the current standard therapy for treatment of hepatitis C viral infection.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history compatible with chronic hepatitis C and compensated liver disease
* Failed response to previous hepatitis C therapy of pegylated interferon/ribavirin

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with hepatitis B or HIV

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Francisco, California
  - Miami, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - New York, New York
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas